CLINICAL TRIAL: NCT04341649
Title: Multi-device Testing for Autonomic Nervous System Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, yilong Wang, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 119209
Record Dates: First submitted 2020-03-25; First posted 2020-04-10 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Vagus Nerve Stimulation
Keywords: Parasympathetic Nervous System; Vagus Nerve Stimulation; Head Massage; Low Laser therapy
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: It is a crossover randomized trial where each participant is exposed to one of the 7 types of intervention, allocated randomly. Up to 20 healthy volunteers will be recruited.
Masking Description: Participants may be aware partially or totally of the nature of the intervention. For instance Manual Head Massage or Helmet Massager cannot be blind. However, for LLT or sham LLT the participants will remain blind. Indeed, Relaxed reading time is known by the participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Head massage by therapist (Active Comparator): Head massage therapist will practice massage covering the scalp, front head, occipital area and neck.
  Interventions: Other: Manual Head Massage
- Helmet massage BREO (Active Comparator): Breo helmet will be installed for massaging the head at different defined places.
  Interventions: Device: BREO Helmet Massager
- Low Laser Therapy (Active Comparator): Laser light can penetrate the skin and stimulate the nervous connections. The investigators will use a laser pen (Min Sheng).
  Interventions: Device: Low Laser Therapy (LLT)
- Sham Low Laser Therapy (Active Comparator): The investigators will use the same laser pen, but without laser beam.
  Interventions: Device: Sham LLT
- TENS ear stimulation (Active Comparator): The investigators will use the (Hwato) device that provides electrical pulse at various frequency and intensity. This TENS device is a prototype modified for ear stimulation.
  Interventions: Device: TENS ear stimulation
- Deep and Slow breathing (Active Comparator): This intervention is guided by an app that leads to a full respiratory.
  Interventions: Behavioral: Deep and Slow breathing
- Relaxed Reading time (Sham Comparator): Participants will read the newspaper in a quiet environment.
  Interventions: Behavioral: Relaxed Reading time

INTERVENTIONS:
Other: Manual Head Massage — Duration 10 minutes.
  Arms: Head massage by therapist
Device: BREO Helmet Massager — Duration 10 minutes.
  Arms: Helmet massage BREO
Device: Low Laser Therapy (LLT) — Duration 7 minutes.
  Arms: Low Laser Therapy
Device: Sham LLT — Duration 7 minutes.
  Arms: Sham Low Laser Therapy
Device: TENS ear stimulation — Duration 7 minutes.
  Arms: TENS ear stimulation
Behavioral: Deep and Slow breathing — A full respiratory cycle of 10 seconds with 5 seconds for inspiration and 5 seconds for expiration.
  Arms: Deep and Slow breathing
Behavioral: Relaxed Reading time — Duration 10 minutes.
  Arms: Relaxed Reading time

SUMMARY:
The Vagus nerve (VN) serve as an "unconscious inner brain" that integrates messages from the body and provides metabolic homeostatic regulation to various organs.In this study the investigators want to compare different ways to stimulate the vagus nerve to assess their respective effects compared to a sham stimulation.

Each participant will be exposed in a random way to 7 different ways to stimulate the VN:

* Manual Head Massage
* Mechanical Head Massager (BREO Inc. Helmet)
* Low laser Therapy (LLT)
* Sham LLT
* Transcutaneous Electrical Nervous Stimulation (TENS) ear stimulation (as testing phase prototype device)
* Deep and slow breathing (as testing intervention based on video app)
* Relaxed reading time (as control situation)

Therefore, within the same design the investigators want to conduct two separate studies that should lead to two separate publications:

* Study 1: comparison of manual head massage to mechanical Helmet massager and relaxed reading
* Study 2: comparison of LLT with sham LLT and relaxed reading

The two other interventions: TENS ear stimulation and Deep and Slow breathing are purely observational to gain knowledge in context of a convenient design.

DETAILED DESCRIPTION:
OBJECTIVES Overall objective is to assess the respective effects of the different ways to stimulate the Vagus Nerve on the Heart Rate Variability (HRV) parameters: High Frequency (HF), Low Frequency (LF), Total Power (TP), Heart rate (HR), and blood pressure (BP).

Specific objectives:

* Comparison of Manual Head Massage to Mechanical Head Massager to Control situation
* Comparison of Low Laser Therapy (LLT) to sham LLT to control situation
* Effects of TENS ear stimulation (descriptive)
* Effects of Deep and Slow breathing (descriptive)

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 20 to 40 in normal context

Exclusion Criteria:

* To have work night shift the night before
* To use certain drugs that affect the ANS (beta blockers, beta stimulant, hypnotic, for instance)
* To be in situation of unusual life stress
* To have a chronic disease that require some daily treatment
* Not to stay in Beijing for the duration of the investigation

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Changes of HRV recording parameters | Changes from baseline HRV parameters at post intervention 15 minutes
  The investigators will use the BIOPAC Machine that captures ECG data, signals were sampled at 500 Hz throughout the testing. Recorded data were reviewed and analyzed using AcqKnowledge software version 4.2. The HRV recording parameters include: (1) Very Low Frequency (VLF) (< 0.04 Hz), (2) Low Frequency (LF) (0.04 - 0.15 Hz), (3) High Frequency (HF) (0.15 to 0.4 Hz), (4) Total Power (TP), which was calculated by summing up all frequency bands, (5) Total Power partial (TPp) (HF + LF), (6) HFnu (normalized unit of HF), (7) Ratio (HF divided by LF).

SECONDARY OUTCOMES:
Change of Blood Pressure (Systolic and Diastolic Blood pressure) | Change from baseline systolic and diastolic blood pressure at post intervention 15 minutes
  Both systolic and diastolic blood pressure will be recorded by an automated monitoring device (OMROM - HEM 7124) at baseline (after the 5 minutes rest) and at the end of the 15 minutes follow-up.
Change of Heart Rate | Change from baseline heart rate at post intervention 15 minutes
  Heart rate will be monitored at the same time of blood pressure
Change of Body Tension | Change from baseline body tension at post intervention 15 minutes
  Body tension is assessed using a a 10-point Likert-scale (the minimum score is 0, and the maximum score is 10)ratings of perceived body tension (BT) as indicator of stress. The highers scores indicate more stress.

CONTACTS AND LOCATIONS:
Overall Officials: Collet Jean-Paul, MD, Phd, Principal Investigator — Advanced Innovation Center for Human Brain Protection
Locations (1):
- Center for Autonomic Evaluation and Brain Plasticity Advanced Innovation Center for Human Brain Protection, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Need to contact the PI (Dr Collet). Dataset will be transferred with respect of the privacy and confidentiality
Supporting Information: Study Protocol
Time Frame: About one month
Access Criteria: Demand from one academic center